CLINICAL TRIAL: NCT00635349
Title: A Comparison of Tramadol/Acetaminophen Tablets Maintenance Versus NSAID Maintenance After Tramadol/Acetaminophen and NSAID Combination Therapy in Knee Osteoarthritis Patients: Multicenter, Randomized, Open Comparative Study
Brief Title: A Comparative Study of Tramadol Hydrochloride Plus Acetaminophen Tablets Maintenance Versus Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) Maintenance in Participants With Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR012964; NCT00635349; ULT-KOR-05
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Osteoarthritis
Keywords: WOMAC; Knee osteoarthritis pain; Pain intensity; Tramadol; Acetaminophen; Meloxicam; Aceclofenac
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Meloxicam; aceclofenac; Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-steroidal Anti-inflammatory Drug (NSAIDs) (Active Comparator): Participants will receive fixed dose combination of tramadol hydrochloride 37.5 milligram (mg) plus acetaminophen 325 mg, 1 to 3 tablets per day along with meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 1 to Day 28. Participants who will have the numeric rating scale score 4 or less on Day 29 will be randomly assigned to the treatment of NSAIDs to receive either meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 29 to Day 85.
  Interventions: Drug: Meloxicam; Drug: Aceclofenac; Drug: Tramadol Hydrochloride Plus Acetaminophen
- Tramadol Hydrochloride Plus Acetaminophen (Experimental): Participants will receive fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day along with meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 1 to Day 28. Participants who will have the numerical rating scale score 4 or less on Day 29 will be randomly assigned to the treatment of fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 or 2 tablets 4 times daily from Day 29 to Day 85 (maximum daily dose will be 8 tablets).
  Interventions: Drug: Meloxicam; Drug: Aceclofenac; Drug: Tramadol Hydrochloride Plus Acetaminophen

INTERVENTIONS:
Drug: Meloxicam — Meloxicam 7.5 mg or 15 mg per day along with fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day from Day 1 to Day 28, and meloxicam 7.5 mg or 15 mg per day from Day 29 to Day 85.
Drug: Aceclofenac — Aceclofenac 100 mg twice a day along with fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day from Day 1 to Day 28, and aceclofenac 100 mg twice a day from Day 29 to Day 85.
Drug: Tramadol Hydrochloride Plus Acetaminophen — Fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day along with NSAIDs (meloxicam [7.5 mg or 15 mg once daily] or aceclofenac [100 mg twice daily]) from Day 1 to Day 28, and fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 or 2 tablets 4 times daily from Day 29 to Day 85 (maximum daily dose will be 8 tablets).

SUMMARY:
The purpose of this study is to compare the effectiveness of tramadol hydrochloride 37.5 milligram (mg) plus acetaminophen 325 mg maintenance with that of non-steroidal anti-inflammatory drugs (NSAIDs) maintenance in participants with knee osteoarthritis (a progressive and degenerative joint disease, in which the joints become painful and stiff) whose pain was relieved after the add-on treatment of tramadol hydrochloride to NSAIDs.

DETAILED DESCRIPTION:
This is a multicenter (when more than one hospital or medical school team work on a medical research study), randomized (the study drug is assigned by chance), open-label (all people know the identity of the intervention), comparative study to compare the efficacy of tramadol hydrochloride plus acetaminophen maintenance with that of NSAIDs maintenance in participants whose pain was relieved after the add-on treatment of tramadol 37.5 milligram (mg) plus acetaminophen 325 mg to NSAIDs. All participants will receive tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day along with NSAIDs (meloxicam [7.5 mg or 15 mg once daily] or aceclofenac [100 mg twice daily]) from Day 1 to Day 28, and participants will be randomly assigned into 2 treatment groups at Day 29 if the numerical rating scale score less than or equal 4. Tramadol plus acetaminophen group will receive 1 or 2 tablets containing tramadol 37.5 mg plus acetaminophen 325 mg 4 times daily (maximum daily dose will be 8 tablets) from Day 29 to Day 85 and NSAIDs group will receive either meloxicam 7.5 mg or 15 mg per day or aceclofenac 100 mg twice a day from Day 29 to Day 85. The efficacy will be evaluated on Day 1, Day 29, Day 57 and Day 85. The primary efficacy end point will be assessed through change in Western Ontario McMaster Universities Osteoarthritis Index (WOMAC) total score from Day 29 to Day 85. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have suffered from knee osteoarthritis at least for one year and meet the criteria of American College of Rheumatology
* Participants who are taking stable dose of meloxicam 7.5 milligram (mg) or 15 mg daily or aceclofenac 100 mg twice a day at least for four weeks
* Participants whose mean pain intensity has been 5 or higher on the numeric rating scale (NRS) for the last 48 hours
* Participants whose general health conditions are favorable, according to the criteria below: Medical and medication history, Physical examination before the study medication administration, Vital signs: Blood pressure, pulse, Clinical laboratory tests: Serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvate transaminase (SGPT) less-than or equal to (=<) 2 X normal range, Renal function: Creatinine less than (<) 2.0 milligrams per deciliter (mg/dl)
* Female participants of childbearing potential to use the proper contraceptive methods during the study period (Urine pregnancy test prior to the study participation should be negative)

Exclusion Criteria:

* Participants who are applicable to Kellgren and Lawrence grade
* Participants who had failed tramadol treatment before or stopped taking tramadol due to adverse event(s)
* Participants who are applicable to one of the following conditions: Rheumatoid arthritis, Ankylosing spondylitis, Active gout or active pseudo-gout, Diagnosis of fibromyalgia (according to ACR Criteria), Anserine bursitis, Major trauma of the target joint within six months prior to the study medication administration, Infection of the target joint within six months prior to the study medication administration, Apparent avascular necrosis of the target joint within six months prior to the study medication administration, Anatomical deformities of the target joint, which may interfere with assessment of the target joint, Surgical procedures associated with the target joint within one year prior to the study medication administration, Arthroscopic procedures associated with the target joint within six months prior to the study medication administration
* Participants who have one of the following diseases: Significantly unstable diseases such as sleep disorder (e.g., sleep apnea or narcolepsy) or dementia, Functional damage or disease which may cause malabsorption, excessive accumulation, or metabolism or excretion disorder
* Participants who are pregnant or breast-feeding

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2007-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 143 participants were given informed consent, out of which 3 participants had screening failure.
Groups:
- Non-steroidal Anti-inflammatory Drugs (NSAIDs): Participants received fixed dose combination of tramadol hydrochloride 37.5 milligram (mg) plus acetaminophen 325 mg, 1 to 3 tablets per day along with meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 1 to Day 28. Participants who had the numeric rating scale score 4 or less on Day 29 were randomly assigned to the treatment of NSAIDs either meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 29 to Day 85.
- Tramadol Hydrochloride Plus Acetaminophen: Participants received fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day along with meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 1 to Day 28. Participants who had the numeric rating scale score 4 or less on Day 29 were randomly assigned to the treatment of fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 or 2 tablets 4 times daily from Day 29 to Day 85 (maximum daily dose was 8 tablets).
Period: Overall Study
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Started | 73 | 67
Completed | 29 | 19
Not Completed | 44 | 48
Not completed — Other | 8 | 6
Not completed — Protocol Violation | 18 | 22
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Lost to Follow-up | 4 | 3
Not completed — Adverse Event | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen | Total
Number analyzed (Participants) | 73 | 67 | 140
Age Continuous [Mean (Standard Deviation); unit: years] | 60.0 (8.0) | 62.3 (7.6) | 61.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 56 | 118
  Male | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Day 29 in Western Ontario and McMaster Universities Arthritis Index (WOMAC) Total Score at Day 85
Description: The WOMAC is a self-administered and health status questionnaire designed to capture elements of pain, stiffness and physical impairment in participants with osteoarthritis. It consists of 24 questions (5 questions about pain, 2 about stiffness and 17 about physical function) scored on a visual analog scale (VAS) of 0 to 10 cm (0 cm=no pain to 10 cm=worse pain). Individual question responses are assigned a score between 0=extreme and 4=none. Maximum scores for each element differ and therefore, scores were normalized. Total normalized score ranges from 0=worst to 100=best.
Time Frame: Day 29 and Day 85
Population: Full analysis set (FAS) population included all randomly assigned participants excluding those who violated the major eligibility criteria or had no data at all after randomization. Last observation carried forward (LOCF) method was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Non-steroidal Anti-inflammatory Drugs (NSAIDs): Participants received fixed dose combination of tramadol hydrochloride 37.5 mg plus acetaminophen 325 mg, 1 to 3 tablets per day along with meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 1 to Day 28. Participants who had the numeric rating scale score 4 or less on Day 29 were randomly assigned to the treatment of NSAIDs either meloxicam (7.5 mg or 15 mg once daily) or aceclofenac (100 mg twice daily) from Day 29 to Day 85.
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 59 | 59
units on a scale
  Day 29 | 33.54 (15.01) | 39.44 (14.17)
  Change at Day 85 | -1.88 (11.07) | -0.07 (13.46)
Statistical Analysis 1: Comparison: Non-steroidal Anti-inflammatory Drugs (NSAIDs) vs Tramadol Hydrochloride Plus Acetaminophen; Test type: Non-Inferiority or Equivalence — Non-inferiority was to be concluded if the lower confidence limit interval was less than -1.0 (1-sided , 97.5% confidence interval); p = 0.4258, t-test, 1 sided; Mean Difference (Final Values) = 1.81, 97.5% CI 1-sided [lower limit -6.31]

2. Secondary Outcome: Change From Day 29 in Pain Intensity Score at Day 85
Description: Pain intensity was evaluated by 11- point numeric rating scale ranging from 0 to 10 where, 0=no pain and 10=pain as bad as you can imagine.
Time Frame: Day 29 and Day 85
Population: Full analysis set (FAS) population included all randomly assigned participants excluding those who violated the major eligibility criteria or had no data at all after randomization. Last observation carried forward (LOCF) method was applied. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 56 | 52
units on a scale
  Day 29 | 3.82 (1.22) | 3.81 (1.03)
  Change at Day 85 | 0.14 (1.76) | 0.83 (2.02)
Statistical Analysis 1: Comparison: Non-steroidal Anti-inflammatory Drugs (NSAIDs) vs Tramadol Hydrochloride Plus Acetaminophen; Test type: Superiority or Other; p = 0.0628, t-test, 1 sided; Mean Difference (Final Values) = -0.68, 97.5% CI 1-sided [lower limit -1.41]

3. Secondary Outcome: Number of Participants With Pain Relief
Description: Pain relief was assessed by using a 6-point scale ranging from -1 to 4 where, -1=pain aggravated, 0=no change, 1=slightly relieved, 2=moderately relieved, 3=considerably relieved, and 4=pain completely disappeared. Participants with pain slightly relieved, moderately relieved and completely disappeared were considered as pain relieved.
Time Frame: Day 29, Day 57 and Day 85
Population: FAS population included all randomly assigned participants excluding those who violated the major eligibility criteria or had no data at all after randomization. Here 'n' signifies number of participants evaluable at each time point for each arm respectively.
Measure: Number; unit: participants
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 59 | 59
participants
  Day 29; Pain relieved (n=56, 52) | 49 | 42
  Day 57; Pain relieved (n=47, 41) | 32 | 28
  Day 85; Pain relieved (n=55, 56) | 42 | 35
Statistical Analysis 1: Comparison: Non-steroidal Anti-inflammatory Drugs (NSAIDs) vs Tramadol Hydrochloride Plus Acetaminophen; Test type: Superiority or Other; p = 0.0131, Fisher Exact — Day 29: p-value was calculated by fisher exact test
Statistical Analysis 2: Comparison: Non-steroidal Anti-inflammatory Drugs (NSAIDs) vs Tramadol Hydrochloride Plus Acetaminophen; Test type: Superiority or Other; p = 0.9834, Chi-squared — Day 57; p-value was calculated by Chi-squared test
Statistical Analysis 3: Comparison: Non-steroidal Anti-inflammatory Drugs (NSAIDs) vs Tramadol Hydrochloride Plus Acetaminophen; Test type: Superiority or Other; p = 0.1131, Chi-squared — Day 85; p-value was calculated by Chi-squared test

4. Secondary Outcome: Number of Participants With Overall Assessment on Study Drug by Participants
Description: Participants' overall assessment on study drug was done by using a 5-point scale ranging from -2 to 2 where, -2= very bad, 1= bad, 0=moderate, 1=good and 2=very good. Study drug refers specifically to the randomized treatment received from Day 29 to Day 85.
Time Frame: Day 85
Population: FAS population included all randomly assigned participants excluding those who violated the major eligibility criteria or had no data at all after randomization. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure
Measure: Number; unit: participants
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 57 | 57
participants
  Very bad | 1 | 1
  Bad | 2 | 11
  Moderate | 21 | 22
  Good | 29 | 21
  Very good | 4 | 2

5. Secondary Outcome: Number of Participants With Overall Assessment on Study Drug by Investigator
Description: Investigator was completed overall assessment on study drug by using a 5-point scale (-2 to 2; where, -2= very bad, 1= bad, 0=moderate, 1=good and 2=very good). Study drug refers specifically to the randomized treatment received from Day 29 to Day 85.
Time Frame: Day 85
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 57 | 57
participants
  Very bad | 1 | 0
  Bad | 1 | 6
  Moderate | 21 | 25
  Good | 31 | 24
  Very good | 3 | 2

6. Secondary Outcome: Number of Participants With Categorical Swelling
Description: Swelling was assessed by using a 4-point scale ranging from 0 to 3 where, 0=no swelling, 1=presence of cross fluctuation of fluid (PCFF), 2=patellar ballotment, and 3=swelling that distort the joint contours (SDJC).
Time Frame: Day 29, Day 57 and Day 85
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 59 | 59
participants
  Day 29; No swelling (n=56, 52) | 52 | 45
  Day 29; PCFF (n=56, 52) | 4 | 7
  Day 57; No swelling (n=47, 41) | 43 | 38
  Day 57; PCFF (n=47, 41) | 4 | 3
  Day 85; No swelling (n=55, 56) | 53 | 46
  Day 85; PCFF (n=55, 56) | 1 | 9
  Day 85; Patellar ballotment (n=55, 56) | 1 | 1

7. Secondary Outcome: Number of Participants With Categorical Tenderness
Description: Tenderness was assessed by using a 4-point scale 0 to 3 where, 0= no tenderness, 1= complaint of tenderness, 2=complaint of tenderness with wincing (CTW), and 3=wincing and attempt to withdraw.
Time Frame: Day 29, Day 57 and Day 85
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Number analyzed (Participants) | 59 | 59
participants
  Day 29; No tenderness(n=56, 52) | 33 | 37
  Day 29; Complaint of tenderness (n=56, 52) | 22 | 14
  Day 29; CTW (n=56, 52) | 0 | 1
  Day 29; Wincing and attempt to withdraw (n=56, 52) | 1 | 0
  Day 57; No tenderness(n=47, 41) | 33 | 30
  Day 57; Complaint of tenderness (n=47, 41) | 14 | 10
  Day 57; CTW (n=47, 41) | 0 | 1
  Day 57; wincing and attempt to withdraw(n=47, 41) | 0 | 0
  Day 85; No tenderness(n=55, 56) | 39 | 44
  Day 85; Complaint of tenderness (n=55, 56) | 15 | 10
  Day 85; CTW (n=55, 56) | 0 | 2
  Day 85; Wincing and attempt to withdraw(n=55, 56) | 1 | 0

ADVERSE EVENTS:
Description: Safety population included all participants who received at least 1 dose study drug and had safety data.
Arm/Group | Non-steroidal Anti-inflammatory Drugs (NSAIDs) | Tramadol Hydrochloride Plus Acetaminophen
Serious Adverse Events (participants affected / at risk) | 1/73 | 0/67
Other Adverse Events (participants affected / at risk) | 17/73 | 12/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-steroidal Anti-inflammatory Drugs (NSAIDs) (N=73) | Tramadol Hydrochloride Plus Acetaminophen (N=67)
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-steroidal Anti-inflammatory Drugs (NSAIDs) (N=73) | Tramadol Hydrochloride Plus Acetaminophen (N=67)
Nausea (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 4
Dizziness (Gastrointestinal disorders) | 6 | 5

LIMITATIONS AND CAVEATS:
There was no wash-out period after Day 28 to show drug efficacy in participants whose pain was already relieved and results were not meet the objective by setting inappropriate non-inferiority limit by applying WOMAC total score in hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is canceled.